CLINICAL TRIAL: NCT02415855
Title: Canadian Pradaxa Acute Stroke Safety Study
Acronym: CPASS
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: CSC2012-01
Record Dates: First submitted 2015-04-09; First posted 2015-04-14 (Estimated); Results first posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Ischemic Attack, Transient; Stroke
MeSH Terms: conditions — Ischemic Attack, Transient; Stroke | interventions — Dabigatran

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Dabigatran
  Other Names: Pradaxa

SUMMARY:
Study Design:

This is a multicentre, prospective, open-label, single arm, phase IV registry study. No additional procedures are included in the study. Standard clinical data will be collected. This will include a physical examination and NIHSS score assessment at baseline. In addition, all neuro-imaging will be collected. Standard imaging includes a non-contrast CT brain at baseline and 7±2 days post-treatment. Repeat NIHSS score assessment at the time of the 7 day CT scan. Repeat clinical and NIHSS score assessment 30 days post-enrolment will also be collected when performed as part of standard care.

Study Objectives:

1. Demonstrate the safety of early dabigatran initiation after minor stroke/TIA in patients with atrial fibrillation.
2. Determine the frequency of asymptomatic hemorrhagic transformation after 7 days of dabigatran treatment following stroke/TIA
3. Determine the effect of asymptomatic hemorrhagic transformation on functional and neurological outcome at 30 days.

DETAILED DESCRIPTION:
Study Aim and Design:

The primary aim of the CPASS registry is to demonstrate the safety of early anticoagulation with dabigatran following cardioembolic stroke. CPASS is a prospective open label single arm observational study. Safety will be established by demonstrating low rates of hemorrhage in this setting.

Administrative Structure:

CPASS is a Canadian Stroke Consortium led study. The study coordinating centre is at the University of Alberta. Case report forms and data monitoring will be completed electronically, using an online EDC system. All imaging data will be read centrally at the Stroke Imaging Laboratory at the University of Alberta.

Study Design Considerations:

A randomized controlled design was considered (dabigatran versus warfarin). This is considered impractical for a number of reasons. Novel oral anticoagulants are recommended as first line agents for stroke prevention in AF patients by the Canadian Cardiovascular Society.19 These agents are associated with improved safety with respect to bleeding complications. This makes randomization of a patient to warfarin who would otherwise be prescribed dabigatran somewhat ethically dubious. In addition, a randomized design would necessitate a very large study, which would not be completed in a reasonable period of time. A registry design allows us to address the question of safety in a systematic fashion. A safety threshold has been defined for any anticoagulant use early after stroke, based on the rates of warfarin-associated intracranial hemorrhage, which have been reported to be 0.5 to 2.5 per 100 patient years.20-24 The registry design therefore permits determination of whether or not dabigatran is within this threshold. Finally, the systematic collection of clinical and imaging data will allow us to determine any risk factors for hemorrhagic transformation associated with early anticoagulation.

Prescribed Study Treatments:

Patients in whom dabigatran is initiated within 14 days of TIA/stroke symptom onset will be included in the registry. Patients will be treated either at a dose of 110 mg BID or 150 mg BID. The dose and timing of initiation of therapy within that 14 day window will be determined by the treating physician. The factors related to physician choice of initiation time (relative to symptom onset) will be recorded.

Visit Schedule / Clinical Data Collection:

Standard clinical assessments and data will be collected. This will include baseline National Institutes of Health Stroke Scale NIHSS, Glasgow Coma Scale (GCS) and vital signs, which will be recorded in a case report form. Stroke risk factors, past medical history and medications, baseline complete blood count, coagulation profile and renal function tests will also be recorded. CHADS2 and CHADSVaSC scores will also be recorded. Clinical endpoints will be ischemic stroke or intracranial hemorrhage within 30 days of anticoagulant initiation. All cerebral ischemic and intracranial hemorrhagic endpoints will be centrally adjudicated from anonymized clinical records, with the intracranial hemorrhages classified as described above. A data collection form will be filled out for each subject at 30 days post-enrolment indicating clinical status and occurrence of outcome events.

ELIGIBILITY:
Inclusion Criteria:

1. All patients will be ≥ 18 years of age.
2. Minor ischemic stroke, defined as NIHSS score ≤ 3. Transient Ischemic Attack (TIA), defined as acute focal neurological deficits, with complete resolution of symptoms within 24 h of onset. In cases where onset time cannot be established, it will be considered to be the time when the patient was last known to be well.
3. Atrial Fibrillation (AF, paroxysmal or persistent). AF must be confirmed with ECG/Holter monitor, or by history All patients prescribed dabigatran according to the Canadian product label by the treating physician following their stroke/TIA. The decision to treat with dabigatran and the timing of the first dose will be determined by the attending physician, independent of the registry. All patients will have a CT scan or MRI, with findings consistent with an ischemic etiology of symptoms.
4. Ability to obtain informed consent obtained from patient or legally authorized representative.

Exclusion Criteria:

1. Acute or chronic renal failure, defined as eGFR <30 ml/min (Cockcroft Gault formula).
2. Known hypersensitivity to dabigatran or any other contraindication to dabigatran therapy, as per Canadian label information.
3. Prior treatment with dabigatran or any other novel oral anticoagulant (including all Factor Xa antagonists). Treatment with warfarin prior to the stroke/TIA is acceptable, but enrolment cannot begin until the INR is ≤1.5.
4. Prior symptomatic ischemic stroke (TIA is not an exclusion criterion)
5. Any significant ongoing systemic bleeding risk, i.e. active GI/GU bleeding or recent major surgery.
6. Clinically significant recent past history or clinical presentation of ICH, subarachnoid haemorrhage (SAH), arterio-venous (AV) malformation, aneurysm, or cerebral neoplasm. At the discretion of each Investigator.
7. Hereditary or acquired hemorrhagic diathesis.
8. Anticipated inability to comply with follow up.
9. Any condition that, in the judgment of the investigator could impose hazards to the patient if study therapy is initiated or affect the participation of the patient in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Minor Stroke (NIHSS Score ≤ 3) and Transient Ischemic Attack Patients ≥ 18 years of age, with a known history of or demonstrated atrial fibrillation (paroxysmal or persistent), who can be treated with dabigatran following stroke.
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2015-03; Primary Completion 2018-03-31 (Actual); Study Completion 2018-05-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - Ottawa Hospital Research Institute, Ottawa, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were approached after the treating physician's decision to treat with dabigatran within 14 days of stroke/TIA, independent of the registry.
Groups:
- Dabigatran 110 mg BID: Participants with an estimated glomerular filtration rate 30-50 ml/min and/or age 80 years received Dabigatran 110 mg twice a day.
- Dabigatran 150mg BID: Participants who were under 80 yrs of age and who had an estimated glomerular filtration rate of greater than 50 ml/min were treated with dabigatran 150mg BID.
Period: Overall Study
Arm/Group | Dabigatran 110 mg BID | Dabigatran 150mg BID
Started | 37 | 64
Completed | 34 | 62
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran 110 mg BID | Dabigatran 150mg BID | Total
Number analyzed (Participants) | 37 | 64 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 30 | 48
  >=65 years | 19 | 34 | 53
Age, Continuous [Mean (Full Range); unit: years] | 72 [60 to 83] | 72 [60 to 83] | 72 [60 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 22 | 35
  Male | 24 | 42 | 66
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 37 | 64 | 101

OUTCOME MEASURES:

1. Primary Outcome: Symptomatic Hemorrhagic Transformation Rate (PH2)
Description: Symptomatic Hemorrhagic Transformation Rate (PH2) associated with clinical deterioration, defined as worsening of NIHSS score of 4 or more points within 30 days of initiating dabigatran therapy.
Time Frame: 30 days post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran 110 mg BID | Dabigatran 150mg BID
Number analyzed (Participants) | 37 | 64
Participants | 0 | 0

2. Secondary Outcome: Any Parenchymal Haemorrhage (PH1 or PH2)
Description: Any parenchymal haemorrhage (PH1 or PH2) on follow-up CT scan at 7±2 days post-enrolment.
Time Frame: 7 days post-enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran 110 mg BID | Dabigatran 150mg BID
Number analyzed (Participants) | 37 | 64
Participants | 3 | 3

3. Secondary Outcome: Symptomatic Hemorrhagic Transformation Rate
Description: Symptomatic hemorrhagic transformation rate (defined as above) in patients treated with warfarin prior to the index stroke/TIA.
Time Frame: 30 days post enrolment
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran 110 mg BID | Dabigatran 150mg BID
Number analyzed (Participants) | 37 | 64
Participants | 0 | 0

4. Secondary Outcome: Recurrent TIA/Ischemic Stroke
Description: Monitoring and documentation of recurrent TIAs or Ischemic Stroke occuring in participants of both arms
Time Frame: 30 days post enrolment
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran 110 mg BID | Dabigatran 150mg BID
Number analyzed (Participants) | 37 | 64
Participants | 2 | 2

5. Secondary Outcome: Systemic Hemorrhagic Complication Rate
Description: Monitoring and documentation of the number of the rate of hemorrhagic complications for participants in either arm of the study.
Time Frame: 30 days post enrolment
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran 110 mg BID | Dabigatran 150mg BID
Number analyzed (Participants) | 37 | 64
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days from start of medication.
Arm/Group | Dabigatran 110 mg BID | Dabigatran 150mg BID
All-Cause Mortality (participants affected / at risk) | 1/37 | 0/64
Serious Adverse Events (participants affected / at risk) | 1/37 | 0/64
Other Adverse Events (participants affected / at risk) | 1/37 | 1/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dabigatran 110 mg BID (N=37) | Dabigatran 150mg BID (N=64)
Recurrent Stroke (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dabigatran 110 mg BID (N=37) | Dabigatran 150mg BID (N=64)
Bleeding per rectum (Endocrine disorders) | 1 (1) | 0 (0)
Sensory loss/Paresthesias, weak arms and headaches (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-29): https://cdn.clinicaltrials.gov/large-docs/55/NCT02415855/Prot_SAP_000.pdf